

# BMT CTN 1101 CLINICALTRIALS.GOV IDENTIFIER: NCT01597778 PATIENT INFORMED CONSENT DONOR INFORMED CONSENT DONOR ASSENT

Version 8.0 January 18, 2017

THIS DOCUMENT IS CONFIDENTIAL AND PRIVILEGED

## APPENDIX B CONSENT FORMS

## PATIENT INFORMED CONSENT DONOR INFORMED CONSENT DONOR ASSENT

#### **Informed Consent to Participate in Research**

A Multi-Center, Phase III, Randomized Trial of Reduced Intensity(RIC)
Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

| Your Name: | |
|---|---|
| Study Title: | A Multi-Center, Phase III, Randomized Trial of Reduced Intensity(RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies |
| Protocol: | BMT CTN #1101 |
| Co-Investigator: | Ephraim Fuchs, M.D. Johns Hopkins University 488 Bunting-Blaustein Cancer Research Building, 1650 Orleans Street Baltimore, MD 21231 Phone: 410- 955-8143 Email: <a href="mailto:fuchsep@jhmi.edu">fuchsep@jhmi.edu</a> |
| Co-Investigator: | Paul O'Donnell, M.D., Ph.D. Massachusetts General Hospital Cancer Center, 55 Fruit St. Boston, MA 02141Phone: 508-693-7430 Email: <a href="mailto:pvodonnell@mgh.harvard.edu">pvodonnell@mgh.harvard.edu</a> |
| Co-Investigator: | Claudio Brunstein, M.D. University of Minnesota Medical Center 420 Delaware Street SE, MMC 286, Minneapolis, MN 55455 Phone: 612-624-5620 Email: <a href="mailto:bruns072@umn.edu">bruns072@umn.edu</a> |
| Transplant Center Investigator: (Insert contact inforn | nation for PI at your site) |
| Sponsor: | The National Institutes of Health (NIH) is sponsoring this study by providing financial support through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN). |

#### 1. Introduction

We invite you to join this clinical trial, also known as a research study. We are doing this research because we want to learn more about reduced-intensity transplants that use a mismatched donor. These results will help us understand if one kind of mismatched donor is better or if there is no difference at all.

This study will take at least 4 years and will include about 400 participants. Your study participation will last for **3 years** after your transplant.

This Consent Form will tell you about the purpose of the study, the possible risks and benefits, other options available to you, and your rights as a participant in the study.

Everyone who takes part in research at [insert facility name] should know that:

- Being in any research study is voluntary.
- You may or may not benefit from being in the study. Knowledge we gain from this study may benefit others.

- If you join the study, you can quit the study at any time.
- If you decide to quit the study, it will not affect your care at [insert name of facility or institution].
- Please ask the study staff questions about anything that you do not understand, or if you would like to have more information.
- You can ask questions now or any time during the study.
- Please take the time you need to talk about the study with your doctor, study staff, and your family and friends. It is your decision to be in the study. If you decide to join, please sign and date the end of the Consent Form.

You and your doctor will discuss other treatment choices if you do not want to participate in this study.

#### 2. Study Background

The National Institutes of Health (NIH), through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN), are providing staff support and money for this research study. The BMT CTN will direct the research study. The BMT CTN and the

NIH will make decisions about how to manage the study.

A stem cell transplant is the only treatment at this time that <u>may</u> cure your disease. An **allogeneic** transplant uses blood-making cells from a family member or an unrelated

donor to remove and replace your abnormal blood cells. Your doctor may recommend that you have a transplant that uses lower amounts of chemotherapy and radiation. This type of transplant is also called a **reduced intensity**, **non-myeloablative**, or "**mini**" transplant. Because of your age or health problems and because you do not have a matched donor, you may have a higher chance of health problems from a standard stem cell transplant that uses high doses of chemotherapy and/or radiation.

Recent studies by the BMT CTN suggest the results are very similar for reduced-intensity transplants when they use either mismatched cord blood or use mismatched bone marrow from a family member.

There is no guarantee or promise that this procedure will be successful.

#### 3. Study Purpose

We are inviting you to take part in this study because you have a cancer of the blood or lymph glands and a stem cell transplant is a treatment option.

Tissue typing shows that you do not have a completely matched donor available in your family. You also do not have a matched donor outside of your family who can donate when you need them to. However, you do have two other donor choices available for a transplant: (1) partially matched units of unrelated cord blood, and (2) a family donor who is a partial match.

We are doing this research to learn more about reduced-intensity transplants that use a mismatched donor. We will use either cord blood from an unrelated donor or bone marrow from a family member, and then compare the transplant results.

These results will help us understand if one kind of mismatched donor is better or if there is no difference at all.

#### 4. Right to Ask Questions and/or Withdraw

You have the right to ask questions about the study at any time. If you have questions about the study or you want to leave the study, please contact:

[insert contact info for site PI]

Being in this study is voluntary. You can choose not to be in this study or leave this study at any time. If you choose not to take

part or leave this study, it will not affect your regular medical care in any way.

Your study doctor and study staff will be available to answer any questions that you may have about taking part in or leaving this study.

#### 5. Study Treatment and Tests

We will check your health before you start treatment, while you receive treatment, and for several years after you finish your treatment.

#### Before You Start Your Treatment

We will ask you to take quality of life surveys. The surveys will ask about:

- o Any side effects of your treatment
- o Any health problems
- How well you can do things that are important to you
- How you relate to other people
- Your feelings.

You may skip any questions you wish.

We will also ask you to provide optional Blood Samples for Future Research (see Section 18: Optional Blood Samples for Future Research).

Randomization

We will use a computer to randomly assign you to 1 of 2 study groups. One group will receive partially matched cord blood from an unrelated donor, and one group will receive bone marrow from a partially matched family member. You will have an equal chance of being placed in either group.

#### **During Your Treatment**

#### Conditioning Regimen Before Transplant (chemotherapy and radiation)

You will be treated with a type of chemotherapy called **fludarabine**, which is given daily for 5 days. If you receive cord blood, you will also be given a type of chemotherapy called **cyclophosphamide** for 1 day. If you receive bone marrow, you will be given cyclophosphamide for 2 days.

After the chemotherapy is completed, you will receive a small dose of radiation to your whole body (**Total Body Irradiation**) in a single dose. The chemotherapy and radiation may cause side effects. Some of these side effects may be life-threatening (see **Section 6: Risks and Discomforts**).

If you receive cord blood, and have not had cytotoxic chemotherapy within the last 3 months or an autologous transplant within the last 2 years, you will receive a slightly higher dose of radiation (300 cGy instead of 200 cGy). This slightly higher dose of radiation has shown hematopoietic recovery is comparable to that seen with low dose radiation for patients who have had chemotherapy in the last 3 months or an autologous transplant in the last 2 years.

#### Reinfusion of Stem Cells (Transplant)

On your transplant day, if you receive cord blood, it will be given to you through your catheter like a blood transfusion. If you receive bone marrow, your family donor will have his or her marrow collected in the operating room. The donated marrow may be taken to a laboratory where red cells will be removed. The donor cells will be given to you through your catheter and will travel to your bone marrow where they will start to make healthy, new blood cells.

If you receive cord blood you will start to take the immune suppressing drugs cyclosporine and mycophenolate mofetil (MMF) for 3 days before transplant. These drugs may help prevent a complication called graft versus host disease (GVHD; see Section 6: Risks and Discomforts).

If you receive bone marrow, you will be given another dose of cyclophosphamide on Days 3 and 4 after your transplant. You will start to take the immune suppressing drugs **tacrolimus** and MMF to help prevent GVHD on Day 5 after your transplant.

In both study groups (partially matched cord blood from an unrelated donor or bone marrow from a partially matched family member), you will continue to take MMF for about 5 weeks and cyclosporine or tacrolimus for up to 6 months.

If you receive cord blood, you will be given **filgrastim (G-CSF)** through your catheter or by injection under your skin beginning on day 1 after your transplant. If you receive bone marrow, you will be given filgrastim (G-CSF) beginning on Day 5 after your transplant. Filgrastim speeds up the recovery of white blood cells. In both study groups, you will receive filgrastim daily until your white blood cells have recovered.

The immune suppressing drugs and filgrastim may cause side effects. These side effects

may be life-threatening (see Section 6: Risks and Discomforts).

If needed, you will receive blood transfusions to maintain normal blood cell levels and antibiotics to treat or prevent infection. You may also receive extra nutrients and pain drugs during or after your transplant. They will be given to you through your catheter.

#### Health Evaluations

We will test (evaluate) your health during the study. These tests and how often they are scheduled are standard care for patients receiving an allogeneic transplant. They would be done even if you were not part of this study. You will be watched closely for any signs and symptoms of GVHD.

#### Health evaluations after treatment:

- 1) Physical exam to assess toxicities, and infections weekly until Day 56 and then at Days 180, 365, and 730.
- 2) Physical exam to assess GVHD weekly until Day 90 and then at Days 180, 365, and 730.

- 3) Routine blood tests (cell counts and liver and kidney function) weekly until Day 56 and then at Days 180, 365, and 730.
- 4) Blood or bone marrow tests to find the amount of donor cells in your body on Days 28 and 56. This is also called *chimerism*.
- 5) Restaging tests to see how much cancer you have after treatment on Day 730.
- 6) A quality of life survey (see <u>Before You Start Your Treatment</u>) at Days 365 and 730.
- 7) Optional blood samples for future research (see Section 19: Blood Samples for Future Research).

#### Long-term follow-up

Data regarding your clinical situation after 2 years may be obtained from the CIBMTR, which captures information on all US transplants.

#### 6. Risks and Discomforts

You will have side effects while on the study. Side effects can range from mild to very serious.

The risks and discomforts in participating in this study will be similar to what you may have with blood or marrow cell transplant if you do not participate in this trial. Other complications from transplants, such as graft-versus-host disease (GVHD) and infections happen equally in patients who have either type of regimen.

Your health care team will give you medicines to help lower side effects such as feeling sick to your stomach (nausea). In some cases, side effects can be long lasting or may never go away.

#### Risks Related to Medications or Total Body Irradiation Used in Conditioning Regimens

All chemotherapy and radiation treatments used as conditioning regimens in this study

are commonly used in allogeneic hematopoietic cell transplantation.

**TABLE 1 – Risks and Side Effects** 

| Likely | What it means: This type of side effect is expected to occur in more than 20% of patients. This means that 21 or more patients out of 100 might get this side effect. |
|---|---|
| Less Likely | What it means: This type of side effect is expected to occur in 20% of patients or fewer. This means that 20 patients or fewer out of 100 might get this side effect. |
| Rare, but<br>Serious | What it means: This type of side effect does not occur very often – in fewer than 2% of patients – but is serious when it occurs. This means that 1 or 2 patients (or fewer) out of 100 might get this side effect. |

#### Cyclophosphamide (Cytoxan®)

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| <ul> <li>Decreased white blood cell count with increased risk of infection</li> <li>Temporary hair loss</li> <li>Nausea</li> <li>Vomiting</li> <li>Loss of appetite</li> <li>Sores in mouth or on lips</li> <li>Diarrhea</li> <li>Stopping of menstrual periods in women</li> <li>Decreased sperm production in men</li> <li>Decreased platelet count (mild) with increased risk of bleeding</li> <li>Blood in urine</li> </ul> | <ul> <li>Anemia</li> <li>Temporary tiredness</li> <li>Damage to the fetus if you become pregnant while taking drug</li> </ul> | <ul> <li>Scarring of lung tissue, with cough and shortness of breath</li> <li>Severe heart muscle injury and death at very high doses</li> <li>New (secondary) cancers</li> </ul> |

#### Fludarabine (Fludara®)

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| <ul> <li>Decreased white blood cell count with risk of infection</li> <li>Decreased platelet count with increased risk of bleeding</li> <li>Anemia</li> <li>Tiredness</li> <li>Nausea</li> </ul> | <ul> <li>Diarrhea</li> <li>Numbness and tingling in hands and/or feet related to irritation of nerves of the hand and/or feet</li> <li>Changes in vision</li> </ul> | <ul> <li>Pneumonia</li> <li>Agitation or nervousness</li> <li>Confusion</li> <li>Cough</li> <li>Difficulty breathing</li> <li>Weakness</li> </ul> |
| ■ Vomiting | | <ul><li>Severe brain injury and death</li></ul> |

#### Filgrastim (G-CSF; Neupogen®)

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| <ul> <li>Ache or pain inside the bones</li> <li>Increased levels of liver enzymes and uric acid in the blood</li> <li>Low number of platelets in the blood</li> <li>Headache</li> <li>Tiredness</li> </ul> | <ul> <li>Local irritation (skin) at the injection site</li> <li>Nausea</li> </ul> | <ul> <li>Allergic reaction</li> <li>Low fever</li> <li>Enlargement or rupture of the spleen</li> <li>Worsening of preexisting skin rashes</li> </ul> |

#### Mycophenolate mofetil (MMF; CellCept®)

#### **Total Body Irradiation**

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| ■ Fatigue | <ul><li>Vomiting</li></ul> | <ul> <li>Diarrhea</li> </ul> |
| <ul><li>Hair loss</li></ul> | <ul><li>Cataracts</li></ul> | <ul><li>Lung fibrosis</li></ul> |
| <ul><li>Infertility</li></ul> | <ul> <li>Inflammation of the parotid glands</li> </ul> | <ul><li>Second</li></ul> |
| ■ Loss of | <ul> <li>Skin pigmentation (reversible)</li> </ul> | cancers |
| appetite | <ul> <li>Stunted Growth</li> </ul> | |
| <ul><li>Mouth sores</li></ul> | <ul> <li>Low white blood cell count with increased risk</li> </ul> | |
| <ul><li>Nausea</li></ul> | of infection | |
| | <ul> <li>Low platelet count with increased risk of<br/>bleeding</li> </ul> | |
| | <ul><li>Anemia</li></ul> | |

#### Tacrolimus (Prograf®; FK-506)/Cyclosporine

| Likely | Less Likely | Rare, but Serious |
|---|---|---|
| <ul><li>Kidney problems</li></ul> | <ul><li>Nausea</li></ul> | <ul><li>Seizures</li></ul> |
| • Loss of magnesium, calcium, | <ul><li>Vomiting</li></ul> | <ul><li>Changes in vision</li></ul> |
| potassium | <ul><li>Liver problems</li></ul> | <ul><li>Dizziness</li></ul> |
| <ul> <li>High blood pressure</li> </ul> | <ul><li>Changes in how</li></ul> | ■ Red blood cell |
| <ul><li>Tremors</li></ul> | clearly one can | destruction |
| <ul> <li>Increases in cholesterol and</li> </ul> | think | |
| triglyceride | <ul><li>Insomnia</li></ul> | |
| | <ul><li>Unwanted hair growth</li></ul> | |
| | <ul><li>Confusion</li></ul> | |

It is very important that you do not eat grapefruit or drink grapefruit juice while taking Tacrolimus. Grapefruit has an ingredient called bergamottin, which can affect some of the treatment drugs used in this study. Common soft drinks that have bergamottin are *Fresca*, *Squirt*, and *Sunny Delight*.

#### Risks and Toxicities Related to Transplant

The following problems may occur as a result of cord blood or marrow transplant. These risks may occur whether a transplant was done as part of the study or not:

- 1. Slow recovery of blood counts. The red blood cells, white blood cells, and platelets can be slow to recover after blood or marrow transplant. Until your blood counts recover, you will need blood and platelet transfusions, and will be at risk for bleeding and infections. To speed the recovery of the white cells as much as possible you will receive Filgrastim.
- 2. Graft failure. The cord blood or bone marrow stem cells (the "graft") may fail to grow inside your body. Past experience suggests that there can be up to a 10-15% chance of graft failure. If graft failure occurs, this may result in low blood counts for a long period of time. If your counts do not recover, you may need to receive a second transplant. Graft failure can be fatal.
- 3. Graft-Versus-Host Disease (GVHD). GVHD results from the bone marrow or cord blood cells in the graft recognizing your body as foreign and attacking it. In most cases, GVHD can be successfully treated. Sometimes GVHD is severe or difficult to treat and may lead to death. You will be watched closely for this complication and given drugs to prevent and/or treat it.

Acute GVHD may produce skin rash, nausea, vomiting, diarrhea, abdominal pain, abnormalities of liver function, and an increased risk of infection. Chronic GVHD may produce skin rashes, hair loss, thickened dry skin, dry eyes, dry mouth, liver disease, weight loss, diarrhea, and an increased risk of infection. To confirm the diagnosis of acute

or chronic GVHD, you may be asked to have a biopsy (a small sample of your tissue to look at under the microscope) of your skin, gut, or, rarely, your liver.

- **4. Other complications.** Other complications may include:
- a. Damage to the vital organs in your body. The transplant could cause problems in any body organ such as the heart, lungs, liver, gut, kidneys and bladder, or brain. The kidneys and the liver are most likely to be damaged. Some patients will experience serious lung problems from infections or the chemotherapy and radiation.
- b. Serious infections. Full and complete recovery of your immune system may take many months. During this time, there is an increased risk of infections. You will be prescribed certain drugs to reduce the chance of those infections. However, these treatments do not always work. If you have an infection, you may have to stay in the hospital longer or be re-hospitalized after transplant. Although most infections can be successfully treated, some infections may result in death.
- c. Relapse of disease or a new blood cancer. Your leukemia or lymphoma may come back even if the transplant is initially successful. In rare cases, a new blood cancer may develop from the donor cells. Cyclophosphamide can cause damage to blood cells, which may result in a blood cancer such as myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML). The blood cancer usually develops 2-10 years after treatment, or 6 years on average.

The risk of developing a new blood

cancer after allogeneic blood or marrow transplant is probably less than 2%. However, if you receive bone marrow, your donor's marrow is exposed to the chemotherapy drug, cyclophosphamide, after the transplant. There is a risk that a blood cancer may develop in your donor's blood cells. This risk is unknown, but it may be as high as 5%. If cancer develops in your donor's blood cells, you may require additional treatment with chemotherapy or another blood or marrow transplant.

- d. Risk to the unborn. The treatments in this study have <u>not</u> been proven to be safe at any stage of pregnancy. Therefore, if you are pregnant or nursing, you are not eligible for this study. Women who can become pregnant must refrain from all acts of vaginal sex (abstinence) or use two forms of effective birth control while receiving chemotherapy, TBI, and drugs to prevent GVHD. Effective birth control is defined as the following:
  - 1. Consistent use of birth control pills
  - 2. Injectable birth control methods (Depo-Provera, Norplant)
  - 3. Tubal sterilization or male partner who has undergone a vasectomy
  - 4. Placement of an IUD (intrauterine device)
  - 5. Use of a diaphragm with contraceptive jelly and/or condoms with contraceptive foam every time you have sex.

#### Reproductive Risks

The drugs used in this research study may damage your reproductive organs, affect your ability to have children or possibly cause birth defects if you take them while you are pregnant. It is important that a woman is not pregnant or breast-feeding and does not become pregnant during the course of the study.

If you are a woman and can become pregnant, you will need to take a pregnancy test before you start the study. You should discuss ways to prevent pregnancy while you are in the study. Women who have gone through puberty may find that their menstrual cycle becomes irregular or stops permanently. This does not mean that you cannot become pregnant. You must still use two effective methods of birth control or abstinence during your transplant and continue until you are finished with your GVHD prevention treatment.

If you are a man, your body may not be able to produce sperm (become sterile). You should talk with your doctor about banking your sperm before having a transplant.

Please check with your doctor to understand more about these risks.

#### Unforeseen Risks

New risks might appear at any time during the study. These risks might be different from what is listed in this Consent Form. We will promptly tell you about new information that may affect your decision to take part in the study. We may learn new things about reduced-intensity transplants that might make you want to stop being in the study. We will let you know if this happens and you can decide if you want to continue in the study.

#### Additional Information about MMF

- MMF could be damaging to an unborn baby if you are pregnant or become pregnant while receiving the drug.
- MMF can make birth control pills less effective and increase your chances of becoming pregnant while you are taking it.
- If you could become pregnant, you must use 2 effective forms of birth control or abstinence for 4 weeks before starting MMF, during treatment, and for 6 weeks after stopping MMF.
- In this study, you will be assigned to receive MMF for about 5 weeks, so you should not become pregnant during that time. If you think you might be pregnant

or could be become pregnant during the upcoming 5 weeks, you should not join the study.

#### Other Treatments or Drugs

Some drugs react with each other. It is important to tell the study doctor or staff about any other drugs or treatments you are taking. This includes over-the-counter drugs, vitamins and herbal treatments.

It is also important that you tell the study staff about changes to any of your drugs during the study.

For more information about risks and side effects, ask your study doctor.

#### 7. Alternative Treatments

Participation in this study is optional. If you choose not to take part, you may still receive an allogeneic transplant to treat your disease. The treatment and evaluations you would receive could be very similar to what would receive if you join this study.

Your study doctor will talk with you about your options. If you decide not to participate in this study, your medical care will not be affected in any way.

Your other choices may include:

 Treatment with other drugs, radiation, or a combination of drugs and radiation without a transplant

- An allogeneic blood or marrow transplant that is not part of the study, or another type of transplant
- Participation in another clinical trial, if available (check with your doctor)
- No treatment for your blood cancer at this time
- Comfort care

Every treatment option has benefits and risks. Talk with your doctor about your treatment choices before you decide if you will take part in this study.

#### 8. Possible Benefits

Taking part in this study may or may not make your health better. The information from this study will help doctors learn more about reduced-intensity transplant as a treatment for people with a blood cancer and

who have a mismatched donor. This information could help people with a blood cancer who may need a transplant in the future.

#### 9. New Information Available During the Study

During this study, the study doctors may learn new information about the study drug or the risks and benefits of the study. If this happens, they will tell you about the new information. The new information may mean that you can no longer take part in the study, or that you may not want to continue in the study. If this happens, the study doctor will stop your participation and will offer you all available care to meet your needs and medical conditions.

#### 10. Privacy, Confidentiality and Use of Information

Your confidentiality is one of our main concerns. We will do our best to make sure that the personal information in your medical record is kept private. However, we cannot guarantee total privacy. All your medical and demographic (such as race and ethnicity, gender and household income) information will be kept private and confidential. (Name of Transplant Center) and the organizations listed below will not disclose your participation by any means of communication to any person or organization, except by your written request,

or permission, or unless required by federal, state or local laws, or regulatory agencies.

Individuals authorized by the organizations below will have access to your research and medical information. They may use this information for inspections or audits to study the outcomes of your treatment. In agreeing to participate, you consent to such inspections and to the copying of parts of your records, if required by these organizations.

We may give out your personal information if required by law. If information from this

study is published or presented at scientific meetings, your name and other personal information will not be used.

Information about your transplant from your original medical records may be seen or sent to national and international transplant registries, including:

- /Institution/
- The National Institutes of Health (NIH)
- The National Heart, Lung, and Blood Institute (NHLBI)
- The National Cancer Institute (NCI)
- Office of Human Research Protection (OHRP)
- The Food and Drug Administration (FDA)
- Institutional Review Boards (IRBs) responsible for this study

- Data and Safety Monitoring Board (DSMB), not part of /Institution/
- Blood and Marrow Transplant Clinical Trials Network (BMT CTN), including the Center for International Blood and Marrow Transplant Research (CIBMTR), the National Marrow Donor Program (NMDP) and the EMMES Corporation who are coordinating the studies of the BMT CTN
- Study investigators

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

For questions about access to your medical records, please contact /name/ at /number.

#### 11. Ending Your Participation

The study doctor or the study sponsor may stop the study at any time, and we may ask you to leave the study. If we ask you to leave the study, the reasons will be discussed with you. Possible reasons to end your participation in this study include:

- You do not meet the study requirements.
- You need a medical treatment not allowed in this study.

- The study doctor decides that it would be harmful to you to stay in the study.
- You are having serious side effects.
- You become pregnant.
- You cannot keep appointments or take study drugs as directed.
- The study is stopped for any reason.

You could have serious health risks if you stop treatment during the conditioning process before you receive your transplant. If you stop taking the immune suppressing drugs (see **Section 6: Risks and Discomforts**) too soon after transplant, your body could reject the donor stem cells or you could develop serious complications and possibly die.

We ask that you talk with the research doctor and your regular doctor before you leave the study. Your doctors will tell you how to stop safely and talk with you about other treatment choices.

If you decide to leave this study after the start of treatment, or your doctor asks you to leave the study for medical reasons, you will need to come back to the doctor's office for tests for your safety. Even if you leave the study, the information collected from your participation will be included in the study results, unless you specifically ask that it not be included.

#### 12. Physical Injury as a Result of Participation

You will get all available medical treatment if you are injured from taking part in this

study. You and/or your health plan will be charged for this treatment. The study will not pay for medical treatment.

In case you are injured in this study, you do not lose any of your legal rights to receive payment by signing this Consent Form.

#### 13. Compensation or Payment

You will not be paid for taking part in this study. You will not be compensated or reimbursed for any extra costs (for example,

travel and meals) from taking part in this study.

#### 14. Costs and Reimbursements

Most of the visits for this study are standard medical care for your allogeneic transplant and will be billed to your insurance company. You and/or your health plan/insurance company will need to pay for the costs of standard treatment in this study.

Some health plans will not pay these costs for people taking part in studies. Check with your health plan or insurance company to find out if they will pay.

You or your insurance will <u>not</u> be charged for tests that are only done for research on this study.

For questions about your costs, financial responsibilities, and/or medical insurance coverage for your transplant and this study, please contact /Center/ Financial Counselor at /Number/.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Web site at <a href="http://cancer.gov/clinicaltrials/understanding/insurance-coverage">http://cancer.gov/clinicaltrials/understanding/insurance-coverage</a>. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Web site.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

#### 15. For More Information

If you need more information about this study, or if you have problems while taking part in this study, you can contact the study doctor or his/her staff. They can be reached at the telephone numbers listed here:

[Insert name and contact detail]

#### 16. Contact Someone about Your Rights

If you wish to speak to someone not directly involved in the study, or if you have any complaints about the project, or any questions about your rights as a research participant, then you may contact:

[Insert appropriate contact details]

The ethical aspects of this research study have been reviewed and approved by [name of IRB].

For questions about your rights while taking part in this study, call the \_\_\_\_\_\_ [name of center] Institutional Review Board (a group of people who review the research to protect your rights) at \_\_\_\_\_ (telephone number).

#### 17. Cost-effectiveness Research

**Study purpose:** The study doctors want to learn more about the costs of the two types of transplant that are being tested in the larger transplant study: 1) partially matched units of unrelated cord blood and 2) family donors who are a partial match. This research will help doctors know which type of transplant is more cost effective.

**Lead study doctor:** Scott Ramsey of the Fred Hutchinson Cancer Research Center in Seattle is the lead study doctor for the cost-

effectiveness research. Dr. Ramsey is a medical doctor and well-known health economist.

Your health insurance and out-of-pocket medical costs: If you agree to join this study, we will ask for the following information about your health insurance:

- 1) Type
- 2) Provider

- 3) Policy number
- 4) Group number
- 5) Policy holder's name and date of birth

We will also want to know about your out-of-pocket transplant costs (costs not covered by your insurance). The out-of-pocket costs you and your family have to cover are important in understanding the overall cost of transplant, so we want to collect information this information as well. For example, we want to know how much you spend on:

- 1) Medical costs (for example, co-pays, prescriptions)
- 2) Travel and lodging
- 3) Cost of time away from work for both you and your caregivers (family and friends).

Your health insurance and out-of-pocket information is called the 'study data' in this consent form.

How we will use your health insurance information: After you have finished the transplant study, we will use your insurance information to learn about the reimbursements your health insurer made and calculate the cost of your transplant. Illness and transplant-related costs happen before the transplant and go on for many years after, so we want to collect reimbursement information for the 12 months before your transplant, and for the 2 years following.

**Privacy, confidentiality and use of information:** Only the study doctors at the Fred Hutchinson Cancer Research Center will have access to your health insurance and

out-of-pocket cost information (study data). To maintain your confidentiality, we will not link your name to the study data. Also, all of the study doctors signed a confidentiality agreement and promised to keep electronic data protected under passwords and physical data (paper or other media such as CDs) in secure facilities (for example, on-campus locked offices and locked filing cabinets).

Collecting the study data: We will collect your health insurance and out-of-pocket information using an online questionnaire and diary. You will get a user ID number and password to log on to the system. The system was designed to be very user friendly, but we will help you with the online questionnaire and diary over the phone if needed. We will also send email reminders. The option to complete a mail-out survey will also be available.

As stated above, <u>we will collect</u> reimbursement information starting 12 months before your transplant until 2 years after.

We will collect out-of-pocket costs 1 month after your transplant, and again 4 and 7 months after your transplant date. We think each online entry will take between 5 and 25 minutes, but this depends on how much information there is to enter.

Help from your caregiver(s): We ask that you give us the name(s) and contact information of your main caregiver(s). This may be your spouse, partner, parent, adult child or sibling, and friends. You may not feel like using the online diary when you're recovering from your transplant, so we ask

that your caregiver(s) help enter this information

We also want to know the time your caregiver(s) spend caring for you after your transplant and the time they spend away from work or school.

Be sure to talk to your caregiver(s) about this study and get their permission before giving us their name and contact information. If you give us the name of your caregiver(s), we will explain the study to them and what they would need to do. They will also get their own consent form to participate in this study.

Risks to participating: The risks to participating in the cost-effectiveness study are small. We will make every effort to keep your health insurance and out-of-pocket cost information private. We will only use this data to get reimbursement information. A possible risk is the loss of confidentiality

about your medical information, but the chance of this happening is very small.

**Payment and costs:** You will not get paid for participating in this study. You will not be charged for taking part in this study.

If you provide out-of-pocket costs, we will give you a summary of these costs at the end of the study. This may be helpful information for tax reporting.

#### Right to ask questions and/or withdraw:

You do not have to be part of the costeffectiveness research study. Your involvement is totally voluntary and deciding not to be part of this study will not affect the medical care or services you are receiving. You can also leave the study at any time.

For more information: Jordan Steelquist, Fred Hutchinson Cancer Research Center, Seattle (206)-267-7438 or email:jsteelqu@fredhutch.org.

#### 18. Blood Samples for Research (Optional)

This section of the informed consent form is about future research studies that will use blood samples from people who are taking part in the main study. You may choose to give blood samples for these future research studies if you want to. You can still be a part of the main study even if you say 'no' to give blood samples for future research studies.

There are no major risks associated with drawing blood. Having your blood drawn can be uncomfortable and can sometimes cause a bruise. In rare cases, a blood draw can cause fainting. Only trained people will draw your blood.

If you agree to provide blood samples, here is what will happen:

- a.) We will collect five extra blood samples at the same time you have routine blood tests done. The amount of blood collected from you is about 4 tablespoons (50mL) each time. If you weigh less than 50 kg, the amount of blood collected will be based on your weight (1 mL per kg).
- b.) We will collect samples at five different dates in the study: Prior to transplant, Day 28, Day 56, Day 180, and Day 365.
- c.) The blood samples will be sent to the BMT CTN Repository for processing and storage. A repository is a place that protects, stores and sends out samples for approved research studies. All research samples will be given a bar code that cannot be linked to your name or other identifying information by future researchers testing your samples.
- d.) Samples stored in the Repository will be used mainly by clinicians and researchers in the BMT CTN network. In the future, the unused research samples and clinical information will be made available outside of this network.
- e.) Researchers can apply to study the materials stored in the Repository. The BMT CTN Steering Committee and/or the BMT CTN Executive Committee must approve each request before they will share samples or information with researchers. This is to make sure that the investigators requesting the samples are qualified, and that the research is of high quality.

f.) DNA from your stored blood samples might be used in genome-wide association (GWA) studies for a future project either done or supported by the National Institutes of Health (NIH). Genome-wide association studies are a way for scientists to find genes that have a role in human disease or treatment. Each study can look at hundreds of thousands of genetic changes at the same time

If your coded samples are used in such a study, the researcher is required to add your test results and sample information into a shared, public research database. This public database is called the NIH Genotype and Phenotype Database and it is managed by the National Center for Biotechnology Information (NCBI). The NCBI will never have any information that would identify you, or link you to your information or research samples.

Some general things you should know about letting us store your blood samples for research are:

- We will only store samples from people who give us permission.
- Research is meant to gain knowledge that my help people in the future. You will not get any direct benefit from taking part. Additionally, you or your doctor will not be given results and they will not be added to your medical record.
- A possible risk is the loss of confidentiality about your medical information. We will

use safety measures with both your samples and clinical information to make sure that your personal information will be kept private. The chance that this information will be given to someone else is extremely small.

Your blood will be used only for research and will not be sold. The research done with your blood may help to develop new products in the future. You will not get paid for any samples or for any products that may be developed from current or future research.

## You can change your mind at any time about allowing us to use your samples and health information for research.

We ask that you contact [Principal Investigator] in writing and let him/her know you do not want us to use your research samples or health information for research. His/her mailing address is on the first page of this form. However, samples and information that have already been shared with other researchers cannot be taken back or destroyed.

## Health Insurance Portability and Accountability Act 1 (HIPAA<sup>1</sup>) Authorization to use and disclose research purpose

#### A. Purpose:

As a research participant, I authorize the Principal Investigators and the researcher's staff to use and disclose my individual health information for the purpose of conducting the research study:

A Multi-Center, Phase III, Randomized Trial of Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

## B. Individual Health Information to be Used or Disclosed:

My individual health information that may be used or disclosed to do this research includes:

- Demographic information (for example: date of birth, sex, weight)
- Medical history (for example: diagnosis, complications with prior treatment)
- Findings from physical exams

 Laboratory test results obtained at the time of work up and after transplant (for example: blood tests, biopsy results)

## C. Parties Who May Disclose My Individual Health Information:

The researcher and the researcher's staff may collect my individual health information from:

[List hospitals, clinics or providers from which health care information can be requested]

#### D. Parties Who May Receive or Use My Individual Health Information:

The individual health information disclosed by parties listed in item c and information disclosed by me during the course of the research may be received and used by the following parties:

Principal Investigator and the researcher's staff

#### **Study Sponsors**

- National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI), both of the National Institutes of Health (NIH),
- Blood and Marrow Transplant Clinical Trials Network (BMT CTN), data and coordinating center

<sup>1</sup> HIPAA is the Health Insurance Portability and Accountability Act of 1996, a federal law related to privacy of health information

 U.S. government agencies that are responsible for overseeing research such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP)

U.S. government agencies that are responsible for overseeing public health concerns such as the Centers for Disease Control (CDC) and federal, state and local health departments.

### E. Right to Refuse to Sign this Authorization:

I do not have to sign this Authorization. If I decide not to sign the Authorization, I will not be allowed to participate in this study or receive any treatment related to research that is provided through the study.

My decision not to sign this authorization will not affect any other treatment, payment, or enrollment in health plans or eligibility for benefits.

#### F. Right to Revoke:

I can change my mind and withdraw this authorization at any time by sending a written notice to the Principal Investigator to inform the researcher of my decision.

If I withdraw this authorization, the researcher may only use and disclose the protected health information already collected for this research study. No further health information about me will be collected by or disclosed to the researcher for this study.

#### **G.** Potential for Re-disclosure:

My individual health information disclosed under this authorization may be subject to re-disclosure outside the research study and no longer protected.

Examples include potential disclosures for law enforcement purposes, mandated reporting or abuse or neglect, judicial proceedings, health oversight activities and public health measures.

#### H. Genetic Information Nondiscrimination Act (GINA)

A new federal law (2009), called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and employers of 15 or more persons to discriminate against you based on your genetic information.

Health insurance companies and group health plans may not request your genetic information that we get from this research. This means that they must not use your genetic information when making decisions regarding insurability. Be aware that this new federal law will not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

## I. This authorization does not have an expiration date.

**TITLE:** A Multi-Center, Phase III, Randomized Trial of Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

PROTOCOL NUMBER: BMT CTN #1101

#### **CO-INVESTIGATOR:**

Ephraim Fuchs, M.D. Johns Hopkins University 488 Bunting-Blaustein Cancer Research Bldg 1650 Orleans Street, Baltimore, MD 21231

Phone: 410- 955-8143 Email: <u>fuchsep@jhmi.edu</u>

#### **CO-INVESTIGATOR:**

Claudio Brunstein, M.D. University of Minnesota Medical Center 420 Delaware Street SE, MMC 286 Minneapolis, MN 55455

Phone: 612-624-5620 Email: bruns072@umn.edu

#### **CO-INVESTIGATOR:**

Paul O'Donnell, M.D., Ph.D. Massachusetts General Hospital Cancer Center 55 Fruit St, Boston, MA 02141

Phone: 508-274-7430

Email: pvodonnell@mgh.harvard.edu

I have read and understood this Consent Form. The nature and purpose of the research study has been explained to me.

- I have had the chance to ask questions, and understand the answers I have been given. I understand that I may ask questions at any time during the study.
- I freely agree to be a participant in the study.
- I understand that I may not directly benefit from taking part in the study.
- I understand that, while information gained during the study may be published, I will not be identified and my personal results will stay confidential.
- I have had the chance to discuss my participation in this research study with a family member or friend.
- I understand that I can leave this study at any time, and doing so will not affect my current care or prevent me from receiving future treatment.

| • | I understand that | I will be given | n a copy of this | signed conser | nt form |
|---|---|---|---|---|---|

| Participant Name | Date |
|------------------|------|
| Signature | Date |

B-26

#### **Statement of Consent for Cost Effectiveness Research**

The purpose of the cost effectiveness research, the procedures involved, and the risks and benefits have been explained to me. I have asked all the questions I have at this time and I have been told whom to contact if I have more questions. I have been told that I will be given a signed copy of this consent form to keep.

I understand that I do not have to participate in the cost effectiveness research. If I decide to not

| participate, it will not affect my medical care in ar | ny way. |
|---|---|
| ☐ I agree to be part of the cost-effectiveness resea | rch. |
| ☐ I do not agree to be part of the cost-effectivenes | s research. |
| Signature | Date |
| Statement of Consent for Research Samples The purpose of storing blood samples, the procedu been explained to me. I have asked all the question whom to contact if I have more questions. I have this consent form to keep. | ns I have at this time and I have been told |
| I understand that I do not have to allow the use of you store research samples now or in the future, it | = |
| I voluntarily agree that my blood and information<br>and/or NHLBI Repositories for research to learn a<br>understand that my DNA and clinical information<br>association studies. | bout, prevent, or treat health problems. I also |
| ☐ I agree to allow my blood samples to be stored: | for research. |
| ☐ I do <u>not</u> agree to allow my blood samples to be | stored for research. |
| Signature | Date |
| I certify that I have provided a verbal explanation<br>the procedures and risks. I believe the participant | , |
| Name of Counseling Physician | Date |
| Signature of Counseling Physician | <br>Date |

#### **Donor Informed Consent to Participate in Research**

A Multi-Center, Phase III, Randomized Trial of Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

| Your name: | |
|---|---|
| Study Title: | Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies |
| Protocol: | BMT CTN #1101 |
| Co-Investigator: | Ephraim Fuchs, M.D. Johns Hopkins University 488 Bunting-Blaustein Cancer Research Building, 1650 Orleans Street Baltimore, MD 21231 Phone: 410- 955-8143 Email: fuchsep@jhmi.edu |
| Co-Investigator: | Paul O'Donnell, M.D., Ph.D. Massachusetts General Hospital Cancer Center55 Fruit St, Boston, MA 012141Phone: 508-274-7430Email: <a href="mailto:pvodonnell@mgh.harvard.edu">pvodonnell@mgh.harvard.edu</a> |
| Co-Investigator: | Claudio Brunstein, M.D. University of Minnesota Medical Center 420 Delaware Street SE, MMC 286, Minneapolis, MN 55455 Phone: 612-624-5620 Email: <a href="mailto:bruns072@umn.edu">bruns072@umn.edu</a> |
| Transplant Center Investigator: (Insert contact inform | nation for PI at your site) |

**Sponsor:** The National Institutes of Health (NIH) is sponsoring this study by providing financial support through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN).

#### 1. Introduction

This informed consent form is about future research studies. These studies will use blood and bone marrow samples from people who take part in the main study titled BMT CTN #1101. You must be 18 years of age or older to give bone marrow samples for future research.

You may choose to give blood and marrow samples for these future research studies if you want to. Your family member can still be a part of the main study even if you say 'no' to giving blood and marrow samples for future research

The main study will use either umbilical cord blood (cord blood) from an unrelated donor or bone marrow from a family member (you), and then compare the transplant results. These results will help us understand if one kind of mismatched donor is better or if there is no difference at all.

If you agree to give blood and marrow samples (marrow from donors 18 and older only), we will collect the blood sample at the same time you have routine blood tests done and the marrow sample at the same time you donate marrow. We hope to collect samples from 200 bone marrow donors who are a part of the main BMT CTN #1101 study.

This Consent Form will tell you about the purpose of the samples for future research, the possible risks and benefits, other options available to you, and your rights as a research participant.

Everyone who takes part in research at [insert facility name] should know that:

- Being in any research study is voluntary.
- You will not directly benefit from being in the study. Knowledge we gain from this study may benefit others.
- If you give blood and marrow samples for future research, you can change your mind at any time.
- If you decide to quit the study, it will not affect your care or the care of your family member at [insert name of facility or institution].
- Please ask the study staff questions about anything that you do not understand, or if you would like to have more information.
- You can ask questions now or any time during the study.
- Please take the time you need to talk about the study with your doctor, study staff, and your family and friends. It is your decision to provide blood and marrow samples for future research. If you decide to join, please sign and date the end of the Consent Form.

The National Institutes of Health (NIH), through the Blood and Marrow Transplant Clinical Trials Network (BMT CTN), are giving staff support and money for this research study. The BMT CTN will lead the research study and, along with the NIH, will make decisions about how to manage the study.

We wish to collect blood and marrow samples from donors (marrow from donors

age 18 and older only) to be used in future research. The research that may be done with your blood and marrow is not designed to help you but it may help people who have cancer or other diseases in the future

#### 2. Study Purpose

We are collecting extra blood and marrow samples for future research because we want to learn more about reduced-intensity transplants that use a mismatched donor. Samples may also be used in the future by researchers with the BMT CTN and other organizations

#### 3. Right to Ask Questions and/or Withdraw

You have the right to ask questions about the study at any time. If you have questions about your rights as a participant or you want to leave the study, please contact:

[insert contact info]

Giving blood and marrow samples for future research is voluntary. You can choose not to give samples, or change your mind at any time. If you choose not to take part or change your mind, it will not affect your

donation process or the treatment of your family member in the main study in any way.

If you change your mind, your blood and marrow samples will not be used for other research studies or tested further.

Your study doctor and study staff will be available to answer any questions that you may have about giving samples for future research.

#### 4. Study Treatments and Tests

If you agree to give blood and marrow samples (marrow from donors age 18 and older only), here is what will happen:

- a.) We will collect 1 extra blood sample at the same time you have routine blood tests done. The amount of blood collected from you is about 4 tablespoons (50 mL). If you weigh less than 50 kg, the amount of blood collected will be based on your weight (1 mL per kg).
- b.) If you are age 18 or older, we will also collect up to 1 tablespoon (10 mL) of bone marrow when you donate for your family member. 3-5 mL will be saved for future research.
- c.) The blood and marrow samples will be sent to the BMT CTN Repository for processing and storage. A repository is a place that protects, stores, and sends out samples for approved studies. All samples will be given a unique bar code that cannot be linked to you by researchers testing your samples.
- d.) Samples stored in the Repository will be used mainly by clinicians and researchers in the BMT CTN network. In the future, the unused research samples and clinical data will be made available outside of this network.

- e.) Researchers can apply to study the samples stored in the Repository. The BMT CTN Steering Committee and/or the BMT CTN Executive Committee must approve each request before they will share samples or information with researchers. This is to make sure that the investigators who request the samples are qualified, and that the research is of high quality.
- f.) DNA from your stored samples might be used in genome-wide association (GWA) studies for a future project either done or supported by the NIH. Genome-wide association studies are a way for scientists to find genes that have a role in human disease or treatment. Each study can look at hundreds of thousands of genetic changes at the same time.

If your coded samples are used in such a study, the researcher is required to add your test results and sample information to a shared, public research database. This public database is called the NIH Genotype and Phenotype Database and it is managed by the National Center for Biotechnology Information (NCBI). The NCBI will never have any information that would identify you, or link you to your information or research samples.

#### 5. Risks and Discomforts

There are no major risks to having your blood drawn. It can be uncomfortable to have your blood taken and it can sometimes leave a bruise. In rare cases, you might faint. Only trained people will take your blood.

There is not a major risk to give extra research samples of bone marrow when the samples are collected at the same time you donate bone marrow.

Information about the bone marrow donation process for this study can be found

in a separate consent form. Your transplant doctor or study coordinator will give you a copy of the donation consent form.

The donation consent form has more information about the steps to donate, and the risks and side effects of the donation process. Only trained people will collect your bone marrow.

#### 6. Possible Benefits

You will not directly benefit from taking part in this study. The information from this study will help doctors learn more about reduced-intensity transplant as a treatment for people with a blood cancer and

who have a mismatched donor. This information could help people with blood cancers who may need a transplant in the future.

#### 7. Privacy, Confidentiality and Use of Information

Your confidentiality is one of our main concerns. We will do our best to make sure that the personal information in your medical record is kept private. However, we cannot guarantee total privacy. All your medical and demographic (such as race and

ethnicity, gender and household income) information will be kept private and confidential. (Name of Transplant Center) and the organizations listed below will not disclose your participation by any means of communication to any person or

organization, except by your written request, or permission, or unless required by federal, state or local laws, or regulatory agencies.

Individuals authorized by the organizations below will have access to your research and medical information. They may use this information for inspections or audits to study the outcomes of your treatment. In agreeing to participate, you consent to such inspections and to the copying of parts of your records, if required by these organizations.

We may give out your personal information if required by law. If information from this

study is published or presented at scientific meetings, your name and other personal information will not be used.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

For questions about access to your medical records, please contact /name/ at /number/.

#### 8. Ending Your Participation

The study doctor or the study sponsor may stop the study at any time, and we may ask you to leave the study. We may ask you to leave the study if you do not follow directions or if you suffer from side effects of the blood draw or the marrow collection. The study sponsor may decide to end the study at any time. If we ask you to leave the study, the reasons will be discussed with you.

Possible reasons to end your participation in this study include:

- You do not meet the study requirements.
- You become unable to donate bone marrow to your family member.
- The study is stopped for any reason.

#### 9. Physical Injury as a Result of Participation

| It is important that you tell your doctor, |
|----------------------------------------------|
| [investigator's |
| name(s)] or study staff if you feel that you |
| have been injured because you provided |
| blood and marrow samples for future |
| research. You can tell the doctor in person |
| or call him/her at |
| [telephone number]. |

You will get all available medical treatment if you are injured as a result providing blood

and marrow samples for future research. You, or your health plan, or your family member's health plan will be charged for this treatment. The study will not pay for medical treatment.

In case of injury resulting from this study, you do not lose any of your legal rights to seek payment by signing this Consent Form.

#### 10. Payment and Study Costs

You <u>will not</u> be paid for your participation in the research study or for providing blood and marrow samples for future research. You will not be compensated or reimbursed for any extra costs (for example, travel and meals) from taking part in this study.

The visits to collect these samples are standard for bone marrow donors and will be billed to your family member's insurance company.

Your family member's insurance will not be charged for tests that are only done for

research on this study. The costs of shipping and storing your blood and bone marrow samples will be paid by the BMT CTN.

For questions about your costs, financial responsibilities, and/or medical insurance coverage for your transplant and this study, please contact /Center/ Financial Counselor at /Number/.

#### 11. For More Study Information

If you need more information about providing blood and marrow samples for future research, or if you have problems while you are participating in this study, you can contact the study doctor or his/her staff. They can be reached at the telephone numbers listed here:

[Insert name and contact details].

#### 12. Contact Someone About Your Rights

If you wish to speak to someone not directly involved in the study, if you have any complaints about the project, or would like more information about your rights as a research participant, you may contact:

[Insert appropriate contact details].

The ethical aspects of this research study have been reviewed and approved by [name of IRB].

For more information about your rights about providing blood and marrow samples for future research, call the \_\_\_\_\_\_ [name of center] Institutional Review Board (a group of people who review the research to protect your rights) at \_\_\_\_\_ (telephone number).

## Health Insurance Portability and Accountability Act (HIPAA)<sup>2</sup> Authorization to use and disclose research purpose

#### A. Purpose:

As a research participant, I authorize the Principal Investigators and the researcher's staff to use and disclose my individual health information for the purpose of conducting the research study:

A Multi-Center, Phase III, Randomized Trial of Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

## B. Individual Health Information to be Used or Disclosed:

My individual health information that may be used or disclosed to do this research includes:

- Demographic information (for example: date of birth, sex, weight)
- Medical history (for example: diagnosis, complications with prior treatment)
- Findings from physical exams

 Laboratory test results obtained at the time of work up and after transplant (for example: blood tests, biopsy results)

### C. Parties Who May Disclose My Individual Health Information:

The researcher and the researcher's staff may collect my individual health information from:

[List hospitals, clinics or providers from which health care information can be requested]

## D. Parties Who May Receive or Use My Individual Health Information:

The individual health information disclosed by parties listed in item c and information disclosed by me during the course of the research may be received and used by the following parties:

Principal Investigator and the researcher's staff

#### Study Sponsors

- National Heart, Lung, and Blood Institute (NHLBI) and the National Cancer Institute (NCI), both of the National Institutes of Health (NIH),
- Blood and Marrow Transplant Clinical Trials Network (BMT CTN), data coordinating center

<sup>2</sup> HIPAA is the Health Insurance Portability and Accountability Act of 1996, a federal law related to privacy of health information

 U.S. government agencies that are responsible for overseeing research such as the Food and Drug Administration (FDA) and the Office of Human Research Protections (OHRP)

U.S. government agencies that are responsible for overseeing public health concerns such as the Centers for Disease Control (CDC) and federal, state, and local health departments.

### E. Right to Refuse to Sign this Authorization:

I do not have to sign this Authorization. If I decide not to sign the Authorization, I will not be allowed to participate in this study or receive any treatment related to research that is provided through the study.

My decision not to sign this authorization will not affect any other treatment, payment, or enrollment in health plans or eligibility for benefits.

#### F. Right to Revoke:

I can change my mind and withdraw this authorization at any time by sending a written notice to the Principal Investigator to inform the researcher of my decision.

If I withdraw this authorization, the researcher may only use and disclose the protected health information already collected for this research study. No further health information about me will be collected by or disclosed to the researcher for this study.

#### **G.** Potential for Re-disclosure:

My individual health information disclosed under this authorization may be subject to re-disclosure outside the research study and no longer protected.

Examples include potential disclosures for law enforcement purposes, mandated reporting or abuse or neglect, judicial proceedings, health oversight activities and public health measures.

#### H. Genetic Information Nondiscrimination Act (GINA)

A new federal law (2009), called the Genetic Information Nondiscrimination Act (GINA) generally makes it illegal for health insurance companies, group health plans, and employers of 15 or more persons to discriminate against you based on your genetic information.

Health insurance companies and group health plans may not request your genetic information that we get from this research. This means that they must not use your genetic information when making decisions regarding insurability. Be aware that this new federal law will not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance.

## I. This authorization does not have an expiration date.

**TITLE:** Reduced Intensity (RIC) Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for Patients with Hematologic Malignancies

PROTOCOL NUMBER: BMT CTN #1101

#### **CO-INVESTIGATOR:**

Ephraim Fuchs, M.D.
Johns Hopkins University
488 Bunting-Blaustein Cancer Research Bldg
1650 Orleans Street, Baltimore, MD 21231

Phone: 410- 955-8143 Email: <u>fuchsep@jhmi.edu</u>

#### **CO-INVESTIGATOR:**

Claudio Brunstein, M.D. University of Minnesota Medical Center 420 Delaware Street SE, MMC 286 Minneapolis, MN 55455

Phone: 612-624-5620 Email: bruns072@umn.edu

#### **CO-INVESTIGATOR:**

Paul O'Donnell, M.D., Ph.D. Massachusetts General Hospital Cancer Center

55 Fruit St, Boston MA, 02151

Phone: 508-274-7430

Email: pvodonnell@mgh.harvard.edu

I have read and understood this Consent Form. The nature and purpose of providing blood and marrow samples for future research has been explained to me.

- I have had the chance to ask questions, and understand the answers I have been given. I understand that I may ask questions at any time during the study.
- I freely agree to give blood and marrow samples (marrow samples from donors age 18 and older only) for future research.
- I understand that I may not directly benefit from providing samples for future research.
- I understand that, while information gained during research may be published,

- I will not be identified and my personal results will stay confidential.
- I have had the chance to discuss giving blood and marrow samples for future research with a family member or friend.
- I understand that I can change my mind at any time, and doing so will not affect my current care or prevent me from receiving future treatment.
- I understand that I will be given a copy of this signed consent form.

#### Complete Appropriate Item Below, A or B

| A. Adult Donor's Consent | B. Parent's Permission for Minor Donor |
|---|---|
| I have read the explanation about this study<br>and have been given the opportunity to discuss<br>it and to ask questions. I hereby consent to<br>give blood and marrow samples for this study. | I have read the explanation about this study and have been given the opportunity to discuss it and to ask questions. I hereby give permission for my child to give a blood sample for this study. |
| Signature of Adult Donor & Date Signed | Signature of Parent(s)/Guardian & Date Signed |
| THIS CONSENT DOCUMENT HAS BEEN APPROVED FOR USE FROM THROUGH | If other than parent, specify relationship: |
| Signature of Investigator & Date Signed | Signature of Witness & Date Signed |

#### **Pediatric Assent to Provide Extra Samples for Research**

Study Title: A Multi-Center, Phase III, Randomized Trial of Reduced Intensity(RIC)

Conditioning and Transplantation of Double Unrelated Umbilical Cord Blood (dUCB) versus HLA-Haploidentical Related Bone Marrow for

**Patients with Hematologic Malignancies** 

**Protocol:** BMT CTN 1101

#### A. Why am I here?

Your bone marrow is a match for a person in your family who needs a transplant. Your bone marrow grows inside your bones. It helps your body make blood and keeps you healthy. A transplant will collect some of your marrow and give it to a person who needs it to make new, healthy cells. Your body will make more marrow afterwards.

If you give us your permission, we would like to have an extra sample of your blood. We would collect the extra sample at the same time you have other blood tests done. We want to save the samples and use them for research in the future.

#### B. Why are you collecting an extra sample of blood?

Research with blood samples will help us learn more about transplant and other diseases. We will keep all of the extra samples private and store them in a place called a Repository. Your name will not be on the samples. Doctors and other researchers can ask to use the samples in the Repository as a part of their research.

#### C. What will happen to me?

If you say it is OK for us to collect an extra blood sample for research, we will ask you for:

 An extra blood sample. We would collect the extra sample at the same time as you have other blood tests done.

We will watch you carefully for side effects, fevers, infections or other problems.

#### D. Will it hurt?

When you have your blood taken with a needle, it may feel like a pinch. It will hurt for a minute and sometimes the place where the needle went might be red and sore. You might get a little bruise from the needle but it goes away in a few days.

#### E. Will the study help me?

Giving the blood sample for research will not help you.

#### F. What if I have questions?

You can ask any questions that you have about giving an extra blood sample. If you forget to ask a question and think of it later, you can call [insert office number].

#### G. Do I have to be in this study?

If you do not want to give an extra blood sample, you need to tell us and your parent or guardian. Your doctor will not be angry or upset if you do not want to join. You can still give bone marrow to the person in your family who needs it. They will still get the exact same care.

You can say yes now and change your mind at any time.

Please talk this over with your parents before you decide if you want to give an extra blood sample for research. We will also ask your parents to give their permission for you to give an extra sample for research.

| Writing your name on this page means that you agree to give an extra blood sample and know what will happen to you. If you change your mind, all you have to do is tell the person in charge. You and your parent or guardian will get a copy of this form after you sign it. | |
|---|---|
| Signature of Researcher | Date |